CLINICAL TRIAL: NCT02936193
Title: Laparoscopy-assisted Pylorus-vagus Nerve Preserving Gastrectomy in the Treatment of Early Gastric Cancer: Clinical Outcomes of a Randomised Controlled Trial
Brief Title: Laparoscopy-assisted Pylorus-vagus Nerve Preserving Gastrectomy in the Treatment of Early Gastric Cancer
Acronym: LAPPG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LAPPG
Record Dates: First submitted 2016-10-07; First posted 2016-10-18 (Estimated); Last update posted 2019-11-05 (Actual); Status verified 2019-04

CONDITIONS: Early Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Gastroenterostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pylorus preservation (Experimental): Patients undergo Laparoscopic Gastrectomy with Pylorus-preservation
  Interventions: Procedure: Pylorus preservation
- Distal gastrectomy (Active Comparator): Patients undergo Laparoscopic Gastrectomy procedure detailing in distal gastrectomy with D2 lymphadenectomy
  Interventions: Procedure: Distal gastrectomy

INTERVENTIONS:
Procedure: Pylorus preservation — Patients undergo Laparoscopic Gastrectomy featuring pylorus-preservation
  Other Names: Laparoscopic-assisted pylorus preserving gastrectomy
  Arms: Pylorus preservation
Procedure: Distal gastrectomy — Patients undergo laparoscopic gastrectomy in distal gastric resection with D2 lymphadenectomy
  Other Names: Laparoscopic-assisted distal gastrectomy
  Arms: Distal gastrectomy

SUMMARY:
The safety and efficacy of Laparoscopy-assisted Pylorus-preserving Gastrectomy (LAPPG) for the treatment of early gastric cancer (EGC) remain controversial. The investigators conducted a randomized controlled trial to compare LAPPG and laparoscopic distal gastrectomy with D2 lymph node dissections for EGC.

DETAILED DESCRIPTION:
During the procedure, the distal part of the stomach is resected, but a pyloric cuff 2-3 cm wide is preserved. The right gastric artery and the infrapyloric artery are preserved to maintain the blood supply to the pyloric cuff. In addition, the hepatic and pyloric branches of the vagal nerves are preserved to maintain pyloric function. The celiac branch of the posterior vagal trunk is sometimes preserved. All regional nodes except the suprapyloric nodes (No. 5) should be dissected as in the standard D2 procedure. However, there are technical challenges associated with completing all of these procedures.The five-year survival rate after PPG with modified D2 lymph node dissection ranges from 95% to 98%. This rate is comparable to the five-year survival rate after gastric resection for EGC, which ranges from 90% to 98%. In terms of oncologic safety, PPG seems reasonably safe for EGC when the accuracy of preoperative diagnosis can be assured

ELIGIBILITY:
Inclusion Criteria:

* Age older than 18 and younger than 75 years
* Primary gastric adenocarcinoma confirmed pathologically by endoscopic biopsy
* cT1-2N0-3M0 at preoperative evaluation according to AJCC Cancer Staging Manual, 7th Edition
* Expected curative resection via distal subtotal gastrectomy with D2 lymphadenectomy
* Written informed consent

Exclusion Criteria:

* Pregnant or breast-feeding women
* Severe mental disorder
* Previous upper abdominal surgery (except laparoscopic cholecystectomy)
* Previous gastrectomy, endoscopic mucosal resection, or endoscopic submucosal dissection
* Other malignant disease within the past 5 years
* Previous neoadjuvant chemotherapy or radiotherapy
* Unstable angina, myocardial infarction, or cerebrovascular accident within the past 6 months
* Continuous systematic administration of corticosteroids within 1 month before the study
* Requirement of simultaneous surgery for other diseases
* Emergency surgery due to a complication (bleeding, obstruction, or perforation) caused by gastric cancer

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-11-02 (Actual); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival | 3 years
  It is the time that passes from the first date after treatment and the date on which gastric cancer progresses, as demonstrated by laboratory testing, radiologic testing, or clinically.

SECONDARY OUTCOMES:
Postoperative complications | 30 days
Postoperative mortality | 30 days
3 years overall survival | 3 years

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Ethics Committee of Renji Hospital, School of Medicine,Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - Ethics Committee of Renji Hospital, School of Medicine, Shanghai Jiaotong University, Shanghai

IPD SHARING:
Plan to Share IPD: Undecided